CLINICAL TRIAL: NCT05765305
Title: Letrozole and Chromium
Brief Title: Combined Chromium With Letrozole Versus Letrozole Only in Induction of Ovulation in Patients With Polycystic Ovary Syndrome
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohammed salah Nasr, Clinical professor, Cairo University
Other Study IDs: 505
Record Dates: First submitted 2023-03-01; First posted 2023-03-13 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-02

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Letrozole; Chromium

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Letrozole: Letrozole versus letrozole with chromium
  Interventions: Drug: Letrozole with chromium

INTERVENTIONS:
Drug: Letrozole with chromium — Letrozole versus letrozole with chromium

SUMMARY:
Combined letrozole with chromium versus letrozole only in induction of ovulation in polycystic ovary syndrome

DETAILED DESCRIPTION:
Randomized controlled trial

ELIGIBILITY:
Inclusion Criteria:

* female patients aged from 18 to 35 years Anovulatory cycles Pcos

Exclusion Criteria:

* female patients aged more than 35years Male factor of infertility Other factors of infertility than pcos

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Female patients aged from 18 to 35 years
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Efficacy of letrozole | 12 months
  efficacy of letrozole with chromium in improving induction of ovulation

SECONDARY OUTCOMES:
Miscarriage rate | 12 months
  Incidence of OHSS

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine, Cairo, القاهره, Egypt

IPD SHARING:
Plan to Share IPD: No
Now no plan